CLINICAL TRIAL: NCT05247450
Title: Conventional-therapy & FES-therapy In-Veritas Effects Study (C-FIVE Study): Rehabilitation of the Upper Extremity for New Persistent C5 Palsy After Surgical Treatment of Patients With Degenerative Cervical Myelopathy
Brief Title: Conventional-therapy & FES-therapy In-Veritas Effects Study
Acronym: C-FIVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Unity Health Toronto (Other); Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-5580
Record Dates: First submitted 2021-10-29; First posted 2022-02-18 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: C5 Palsy
Keywords: Functional electrical stimulation therapy; Degenerative Cervical Myelopathy
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FES-t along with conventional physiotherapy (Experimental): Combined conventional physiotherapy and functional electrical stimulation therapy (FES-t) along with task-specific training
  Interventions: Device: Functional electrical stimulation therapy (FES-t); Other: Conventional physiotherapy
- Conventional physiotherapy alone (Active Comparator): Conventional physiotherapy alone (current standard of care)
  Interventions: Other: Conventional physiotherapy

INTERVENTIONS:
Device: Functional electrical stimulation therapy (FES-t) — Functional electrical stimulation therapy (FES-t) that will use a multichannel device (MyndSearch device).
  Arms: FES-t along with conventional physiotherapy
Other: Conventional physiotherapy — Conventional physiotherapy is the current standard of care for rehabilitation of C5 palsy
  Other Names: Standard of Care

SUMMARY:
This randomized clinical trial will primarily compare the effectiveness of conventional physiotherapy alone with combined conventional physiotherapy and FES-t along with task-specific training in terms of the improvement of the functional and neurological recovery of patients with persistent C5 palsy.

DETAILED DESCRIPTION:
This randomized clinical trial will primarily compare the effectiveness of conventionalphysiotherapy alone with combined conventional physiotherapy and FES-t along with task-specific training in terms of the improvement of the functional and neurological recovery of patients with persistent C5 palsy. Secondarily, this clinical trial will evaluate the effectiveness of combined conventional physiotherapy and FES-t along with task-specific training outcome compared to conventional physiotherapy alone with regards to improved connectivity andexcitability in the ascending and descending pathways as assessed using neurophysiological tests and functional MRI analysis.

ELIGIBILITY:
Inclusion Criteria:

* New unilateral or bilateral, persistent C5 palsy (for at least 3 months) after surgical treatment for degenerative cervical myelopathy

Exclusion Criteria:

* Contraindication for FES-t
* Contraindication for neurophysiological testing
* Contraindication for MRI scanning
* Uncontrolled cardiovascular conditions
* Other medical conditions that can limit treatment protocols
* Other neurological diseases
* Significant persisting mental illness
* Diagnosed learning disabilities
* Substance abuse over 6 months prior to recruitment
* Hearing and visual deficits sufficient to affect test performance
* Reduced passive range of motion (ROM) of the shoulder ("frozen shoulder")
* Inability to participate in and intensive outpatient rehabilitation program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-08-16 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Spinal Cord Independence Measure (SCIM) score | up to 10 weeks post-intervention
  The SCIM is a clinician-administered disability scale developed to specifically address the ability of SCI patients to perform basic activities of daily living independently (SCIM varies from 0 (completely dependent) to 100 (completely independent).

SECONDARY OUTCOMES:
Change in Manual muscle testing | up to 10 weeks post-intervention
  Clinical assessment of the muscle power that varies from 0 (complete paralysis) to 5 (normal)
change in Modified Japanese Outcome Association (mJOA) Score | up to 10 weeks post-intervention
  Clinical assessment of the upper and lower extremities, and bladder function (mJOA varies from 0 [most impaired and disabled] to 18 [normal function]).
Change in neurophysiological parameters | up to 10 weeks post-intervention
  Neurophysiological parameters of neuroplasticity
Change in Functional Magnetic Resonance Imaging (MRI) | 6 to10 weeks post-intervention
  Functional MRI analyses will be focused on improvement of the functional connectivity within the somatosensory and motor cortices and pathways in the brain.

CONTACTS AND LOCATIONS:
Overall Officials: Julio C Furlan, MD,PhD, Principal Investigator — KITE-TRI, University Health Network & University of Toronto
Locations (1):
- KITE Toronto Research Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided